CLINICAL TRIAL: NCT02228161
Title: The Effects of Yoga on Work-related Stress and Stress Adaption Among the Professional Helpers of Psychiatry
Brief Title: The Effects of Yoga in Mental Health Professional Helpers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-Hui Yeh, RN, PhD, Professor, Chang Bing Show Chwan Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 101107
Record Dates: First submitted 2014-08-27; First posted 2014-08-28 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Occupation-related Stress Disorder
Keywords: Yoga; Work-related Stress,; Stress Adaptation.
MeSH Terms: conditions — Occupational Stress | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga exercise (Experimental): Participatants will receive regular 60-minutes yoga classes twice a week for 3 months.
  Interventions: Behavioral: Yoga
- Regular schedule of daily living (No Intervention): Participants will maintain regular schedule as usual.

INTERVENTIONS:
Behavioral: Yoga — Yoga group will receive regular 60-minutes yoga classes twice a week for 3 months.
  Arms: Yoga exercise

SUMMARY:
This study will investigate if yoga exercises decrease work-related stress and improve stress adaptation in professional health helpers.

DETAILED DESCRIPTION:
Mental health professional helpers including psychiatrists, nurses, psychologists, social workers and occupational therapists often call upon to maintain a good working attitude and enthusiasm, especially in the face of the evaluators of credential systems as well as supervisors' authorities. The symptoms of work-related stress of professional helpers developed day by days and affected their physical and mental health. Gradually, the professional helpers burned out. Philip Burnard (1991) mentioned professional helpers might self-neglect while helping others. These would lead to over work related stress that directly affects the physical and mental health of the professional helpers, and indirectly affects the organization to take care of the patients and their families.

According to researchers and personal experience, colleagues of mental health care developed work-related stress symptoms, such as insomnia or sleep disorder, the physiological disorders, weight fluctuations, irritable or depressed while taking care of psychiatric patients. They might take tranquilizers in order to maintain the quality of work. On the other hand, in April 2012, the researchers engaged in yoga teaching, assisting mental health care to help others of engaging in yoga practice showed that members perceived positive feelings after the yoga practice: "the mood is more relaxed," "tight body become more relaxed and soft resulting in awareness of tension and unease. This helps to modify long-term adverse stances and reduce body aches and/or sitting." For this reason, researchers began to apply yoga to the release work-related stress and enhance stress adaptation. Professional health helpers look forward to practice yoga exercises to relax work-related stress and improve stress adaptation.

It is a parallel-arm randomized control trial compare the outcome of participants assign to the experimental treatment group (yoga, with 30 participants) with those assign to a control group for 3 months (12 weeks). Experimental group receive regular 60-minutes yoga classes twice a week. We confer the difference of work-related stress relief and stress adaptation and biofeedback improvement after yoga.

ELIGIBILITY:
Inclusion Criteria:

* Mental Health Professional Helpers.
* Without sport training.
* Age 20~60.

Exclusion Criteria:

* Musculoskeletal injury.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Decrease work-related stress and improve stress adaptation. | 3 months intervention
  Work-related stress and stress adaptation will be assessed by questionnaires including personality, work-related stress and stress adaption scale and biofeedback index using heart rate variability at two different times: (1)baseline data: before yoga program ,(2)outcome data:3 months yoga exercise, right after exercise measures post-test.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hui Yeh Yeh, PhD, Study Director — Show Chwan Memorial Hospital & Central Taiwan University of Science and Technology; Shu-Ling Lin, MS, Principal Investigator — Chang Bing Show Chwan Memorial Hospital
Locations (1):
- Division of Core Laboratory; Chang Bing Show Chwan Memorial Hospital, Changhua County, Taiwan